CLINICAL TRIAL: NCT07155668
Title: A Randomized, Open-label Study Evaluating the Safety, Tolerability and Pharmacokinetics of VRDN-003 Administered Subcutaneously in Participants With Thyroid Eye Disease (TED)
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of VRDN-003 in Participants With Thyroid Eye Disease (TED)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRDN-003-304
Record Dates: First submitted 2025-08-07; First posted 2025-09-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the three study arms.
Masking Description: This is an open label study with no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- VRDN-003 every 4 weeks using autoinjector (Experimental): 6 subcutaneous administrations of VRDN-003 [1 loading dose of 600mg and 5 doses of 300mg]
  Interventions: Drug: VRDN-003; Device: Autoinjector
- VRDN-003 every 8 weeks using autoinjector (Experimental): 3 subcutaneous administrations of VRDN-003 [1 loading dose of 600mg and 2 doses of 300mg]
  Interventions: Drug: VRDN-003; Device: Autoinjector
- VRDN-003 every 8 weeks using vial and syringe (Experimental): 3 subcutaneous administrations of VRDN-003 [1 loading dose of 600mg and 2 doses of 300mg]
  Interventions: Drug: VRDN-003

INTERVENTIONS:
Drug: VRDN-003 — VRDN-003 is an investigational, subcutaneously administered, humanized monoclonal antibody directed against the Insulin-like Growth Factor-1 receptor (IGF-1R).
Device: Autoinjector — The autoinjector is a single-dose, disposable, ready-to-use delivery device
  Arms: VRDN-003 every 4 weeks using autoinjector; VRDN-003 every 8 weeks using autoinjector

SUMMARY:
This is a clinical trial assessing the safety, tolerability and pharmacokinetics (PK) of an investigational drug, VRDN-003, in participants with TED (Thyroid Eye Disease)

DETAILED DESCRIPTION:
This is a randomized (meaning participants will be assigned to study arms by chance), open-label (meaning study doctor, participant and the sponsor will know which study arm participant is assigned to), parallel-group study that will enroll participants with TED of any duration. The key objectives of this study are to determine if VRDN-003 is safe and tolerable and to see how the body reacts to VRDN-003 when administered as a series of subcutaneous (SC) injections every 4 weeks or every 8 weeks in participants with TED either via autoinjector or via vial and syringe.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of TED with or without proptosis, with any CAS (0-7) and in the opinion of the Investigator may benefit from VRDN-003
* Not require immediate ophthalmological or orbital surgery in the study eye for any reason
* Must agree to use highly effective contraception as specified in the protocol
* Female TED participants must have a negative serum pregnancy test at screening

Key Exclusion Criteria:

* Must not have received prior treatment with another anti-IGF-1R therapy
* Must not have received systemic corticosteroids for any condition, including TED, or selenium within 2 weeks prior to first dose.
* Must not have received other immunosuppressive drugs for any condition, including TED, or any other therapy for TED, within 12 weeks prior to first dose
* Must not have received an investigational agent/device for any condition, including TED, within 8 weeks or longer (depending on the type of agent/device) prior to first dose
* Must not have received radioactive iodine (RAI) treatment within 8 weeks prior to first dose
* Must not have had previous orbital irradiation or decompression surgery for TED to the study eye's orbit
* Must not have a pre-existing ophthalmic condition in the study eye which in the study doctor's opinion, would interfere with interpretation of study results
* Must not have abnormal hearing test before first dose or history of ear conditions considered significant by study doctor
* Must not have a history of inflammatory bowel disease
* Female TED participants must not be pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event (TEAE) incidence rate | Through Week 24
  Treatment Emergent Adverse Event (TEAE) incidence rate

SECONDARY OUTCOMES:
Pharmacokinetic outcome measures | Through Week 24
  Time of maximum serum concentration (Tmax) of VRDN-003
Pharmacokinetic outcome measures | Through Week 24
  Maximum serum concentration (Cmax) of VRDN-003

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - United Medical Research Institute, Inglewood, California
  - C&A Clinical Trials Corp, Cape Coral, Florida
  - Ilumina Medical Research, Kissimmee, Florida
  - Med-Care Research, Miami, Florida
  - Continental Clinical Research, llc, Miami, Florida
  - Hype Clinical Research, LLC, Miami, Florida
  - Advanced Quality Medical Research, LLC, Orland Park, Illinois
  - Ophthalmic Consultants of Boston, East Weymouth, Massachusetts
  - Fraser Eye Center, Fraser, Michigan
  - Kahana Oculoplastic and Orbital Surgery, Livonia, Michigan
  - Vector Clinical Trials, Sparks, Nevada
  - Baylor College of Medicine, Alkek Eye Center, Houston, Texas
  - Neuro Eye Clinical Trials INC, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided